CLINICAL TRIAL: NCT06729749
Title: Effect of Bioptron on Primary Dysmenorrhea: a Randomized Controlled Trial
Brief Title: Effect of Bioptron on Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Saleh Ahmed Eldeep, Master student at Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005313
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (control group) (Active Comparator): lt will include 28 participants suffering from PD who will take vitamin D (vit D) supplementations for three consecutive menstrual cycles.
  Interventions: Other: Vitamin D
- Group B (study group) (Experimental): lt will include 28 participants suffering from PD who will take vitamin D (vit D) supplementations as in group A in addition to Bioptron for 20 min daily for 7 days before menstrual cycle along with the first three days of menstrual flow for three consecutive menstrual cycles.
  Interventions: Other: Bioptron Pro 1 Class II; Other: Vitamin D

INTERVENTIONS:
Other: Bioptron Pro 1 Class II — Bioptron Pro 1 Class II: Made by Bioptron AG, Wollerau, Switzerland, a device with a floor stand emits a polarized light lamp. The device has an ergonomic table stand that can be combined with a functional floor stand, allowing flexible use in domestic and professional environments. easily adjustable height and head inclination and the ability to rotate the device head up to 360 allow a convenient usage of nearly any position. Treatments can easily be timed by a control panel down to 30 seconds, an integrated distance rod ensures the recommended distance from the skin surface It will be used for the treatment procedures for all participants in group B only with the following parameters, Wavelengths ranging from 480-3400 nm, Degree of polarization >95% (590 - 1550 nm), Specific power density Av. 40 mW/cm2 Light energy per minute av.2.4 J/cm2, Light Intensity per min. 10.000 lux, Weight without stand 3.4 kg and Weight with stand7.8 kg ,Energy consumption in sleep mode0.5
  Arms: Group B (study group)
Other: Vitamin D — All participants in both groups will take this supplements daily for 3 months

SUMMARY:
This study will be conducted to determine the effect of bioptron on PD through the assessment of serum progesterone level, and pain level measured by pressure algometry in addition to evaluation of the symptoms of PD and its effect on girl's quality of life through valid and reliable questionnaires which will be of valuable benefits in the women's health fields.

DETAILED DESCRIPTION:
All females will be randomly divided into two equal groups:

Group A (control group):

lt will include 28 participants suffering from PD taking vitamin D (vitamin D) supplements for three consecutive menstrual cycles.

Group B (study group):

lt will include 28 participants suffering from PD who will take vitamin D (vitamin D) supplementations as in group A in addition to Bioptron for 20 min daily for 7 days before the menstrual cycle along with the first three days of menstrual flow for three consecutive menstrual cycles.

All females will be given a full explanation of the study protocol and a consent form will be signed by each female before entry in the study

ELIGIBILITY:
Inclusion Criteria:

All females will be clinically diagnosed by the gynecologist with primary dysmenorrhea.

* Self-reported history of PD, at least moderate pain due to menstrual cramps (>4 on VAS)
* They have moderate symptoms of PD on the WaILDD questionnaire, (5-12) Teheran et al., 2018).
* Their ages will be ranged from 18-24 years old.
* Their BMI will be less than 30 kg/m².
* Being a virgin.
* Having regular menstruation for the last 6 months (every 28-30 days with no intermittent bleeding).
* Voluntary acceptance to participate in the study.

B) Exclusion Criteria:

Participants will be excluded if they have:

* Musculoskeletal or neurological disorders.
* Patients with a history of phototherapy allergy.
* Professional athletes (Jill et al., 2012).
* Secondary dysmenorrhea pathology such as (endometriosis, fibroids, adenomyosis, and pelvic inflammatory disease)
* Menstrual irregularity.
* Using hormonal contraception (such as contraceptives or injections).

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Three months
  The pain intensity will be assessed through VAS for both groups (A&B) before and after the end of the treatment program (throughout three consecutive menstrual cycle) and follow up period . Each female will be asked to mark a point on the line between the extreme that is related to her pain intensity.
Pressure pain threshold (PPT) | three months
  A pressure algometer will be used to measure pressure pain thresholds for all participants in both groups (A&B) before and after the treatment program (throughout three consecutive menstrual cycles)

SECONDARY OUTCOMES:
Plasma Progesterone level | Three months
  Plasma progesterone for all participants in both groups (A&B )will be analyzed by Enzyme-Linked Immunosorbent Assay (ELISA), using Cayman Chemical Reagent Company kits before and after the treatment program.
Assessment of menstrual symptoms | Three months
  The WaLIDD questionnaire: will be used to assess the symptoms of primary dysmenorrhea for all participants in both groups (A&B) before the treatment and after the end of the treatment program (throughout three consecutive menstrual cycles and during the follow-up period).
Quality of life enjoyment and satisfaction | Three months
  The Quality-of-life enjoyment and satisfaction questionnaire Q-LES-QSF: will be used to assess health-related quality of life for all participants in both groups (A&B) before the treatment program and after the end of the treatment program (throughout three consecutive menstrual cycles).

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Osman, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No